CLINICAL TRIAL: NCT06259383
Title: A Randomized Controlled Trial of Oral Ivermectin for Patients With Chikungunya Viral Infection During Urban Outbreak in Southern Thailand
Brief Title: Oral Ivermectin for Chikungunya Viral Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Sarunyou Chusri, Principal Investigator, Prince of Songkla University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EC:55-141-14-1-3/sub1
Record Dates: First submitted 2024-01-26; First posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Clinical Syndrome
MeSH Terms: interventions — Ivermectin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients received oral ivermectin, adjunctive to conventional treatment (Experimental)
  Interventions: Drug: Ivermectin
- Patients received conventional treatment (No Intervention)

INTERVENTIONS:
Drug: Ivermectin — 3-day 1 daily dose of 400 μg/kg oral ivermectin
  Arms: Patients received oral ivermectin, adjunctive to conventional treatment

SUMMARY:
Chikungunya viral infection (CVI) is a mosquito-borne infection, caused by chikungunya virus (CHIKV), an alphavirus, belonging to the family Togaviridae. This infection causes febrile illness associated with high fever, rash, acute deliberating and persistent arthralgia. There is no licensed vaccine or specific treatment for this infection. Ivermectin (IVM), commonly-used antiparasitic, has been demonstrated to inhibit replication of CHIKV.

ELIGIBILITY:
Inclusion Criteria:

* patients with virologic confirmation of chikungunya infection who had symptoms less than 72 hours prior to visit

Exclusion Criteria:

* patients with virologic confirmation of chikungunya infection who had symptoms more than 72 hours prior to visit

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2024-01-26 (Actual)

PRIMARY OUTCOMES:
Day of fever clearance | 1 week
  120 participants would be under Body Temperature Assessment - the staff would assess once daily until the fever clearance was below 38C and the measure proportion of patients with fever clearance in each day of assessment until fever clearance at least in 7 days

SECONDARY OUTCOMES:
Day of virologic clearance | 1 week
  120 participants would be obtained blood examination for virological testing every day until virological clearance at least in 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Songkla University, Hat Yai, Changwat Songkhla, Thailand

IPD SHARING:
Plan to Share IPD: No